CLINICAL TRIAL: NCT06475001
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, Dose Response Trial With the Full-spectrum Cannabis Extract VER-01 in Patients With Chronic Non-specific Low Back Pain
Brief Title: Dose-Response Characterization of VER-01 in the Treatment of Patients With Chronic Non-specific Low Back Pain
Acronym: RESPONSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VER-CLBP-004; 2023-507358-34 (EudraCT Number); 1008617 (Other: IRAS ID)
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Chronic Pain; Neuropathic Pain; Back Pain; Back Pain, Low; Back Pain Lower Back Chronic
MeSH Terms: conditions — Chronic Pain; Neuralgia; Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomized to one of four different dose groups (cohorts) in a 1:1:1:1 ratio and either active drug (VER-01) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VER-01 (Experimental): VER-01 is administered orally (b.i.d.) using a dosing syringe. One unit corresponds to 2.5 mg THC. The patient is assigned a fixed dose according to their cohort.
  Interventions: Drug: VER-01
- Placebo (Placebo Comparator): Placebo is administered orally (b.i.d.) using a dosing syringe. The patient is assigned a fixed dose according to their cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VER-01 — Herbal medicinal product, containing as active substance a soft extract of Cannabis sativa L., cannabis flos (Cannabis flower), adjusted to a content of 50 mg/g delta-9-tetrahydrocannabinol (THC).
  VER-01 is adjusted to a concentration of 19 mg/mL THC by adding the excipient sesame oil.
  Arms: VER-01
Drug: Placebo — Comparator without active ingredient
  Arms: Placebo

SUMMARY:
Dose-response characterization of VER-01 in patients with chronic non-specific low back pain (CLBP) for whom drug treatment is indicated and previous optimized treatments with non-opioid analgesics have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.

DETAILED DESCRIPTION:
The primary objective of this multicenter, double-blind, randomized, placebo-controlled trial is to characterize the dose-response relationship of VER-01 in terms of pain reduction in patients with chronic non-specific low back pain.

Eligible patients are randomized to one of four different dose groups (cohorts) in a 1:1:1:1 ratio and either active drug (VER-01) or placebo.

The secondary objectives are to evaluate the efficacy using additional outcome measures, the safety and the tolerability of VER-01 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets the Quebec Task Force (QTF) classification system of categories 1 to 3 of low back pain
2. Male and female patients ≥ 18 years of age
3. Provision of informed consent form (ICF) voluntarily signed and dated by the patient
4. For female patients of childbearing potential and male patients of reproductive potential: use of a reliable contraceptive method (Pearl index < 1) at least 1 month before the screening visit and willingness to use it during the trial participation and 3 months after the last intake of the test or comparative intervention
5. Patient understands the local language and is willing and able to comply with scheduled visits, treatment plan, eDiary, and other trial-related procedures throughout trial participation
6. Chronic (≥ 3 months) non-specific pain in the lower back (between the 12th thoracic vertebra and lower gluteal folds). Non-specific pain refers to pain without a clear specific somatic cause, for which targeted therapy can have a positive effect on the course of the disease. Such somatic causes are e.g., herniated vertebral disk, spinal canal stenosis, inflammatory back pain, osteoporosis, fracture, infection, tumor, spondylolisthesis
7. Patients with indicated opioid drug treatment* where previous optimized treatments** with non-opioid analgesics (including combinations) have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance
8. Low back pain intensity on average ≥ 4 points on an 11-point NRS in the last 4 weeks prior Visit 1
9. In case of non-drug therapy in the 4 weeks prior to Visit 1 (e.g., exercise or behavioral therapy, acupuncture, massage, thermotherapy) that significantly modulates pain perception: the non-drug therapy was unchanged and is still ongoing at Visit 1 and all requirements for continuation of the therapy throughout the trial are given (e.g., prescription, patient's compliance). Ongoing non-drug therapies should be continued unchanged during trial participation
10. Willingness to not take or use any prohibited medication during trial participation. The intake or use of any additional analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics and muscle relaxants), during trial participation is prohibited (except rescue medication). Likewise, strong inhibitors, substrates, or inducers of CYP2C9 and CYP3A4 are considered prohibited concomitant medication in this trial

Exclusion Criteria:

1. Patients with a known history of alcohol/drug/medication abuse (except nicotine) or any dependency or addiction (physical or behavioral) and previous or current use of methadone
2. Evidence of drugs of abuse or illegal drugs by urine drug test performed at Visit 1
3. Known intolerance or hypersensitivity to ingredients of rescue medication, VER-01, and/or placebo (e.g., sesame oil)
4. Participation in another clinical interventional trial within the last 30 days prior Visit 1 or previous participation in a trial for VER-01
5. Occupational groups with primary activity of operating machinery and driving motor vehicles
6. Planned blood donation, planned pregnancy, or planned donation or freezing of sperm or oocytes during trial participation and 3 months after end of trial participation
7. Pregnant or breastfeeding female patients
8. Patient is unable to provide written informed consent, in need for care, has a guardian/caretaker, is immobile, or is particularly vulnerable (e.g., imprisoned; institutionalized by an administrative or judicial authority; dependent or employed by the Sponsor, an external service provider of the Sponsor (involved in the conduct of the trial), the investigator, or the trial site)
9. Known use of THC-containing drugs within 30 days prior Visit 1
10. Patients deemed non-responsive to cannabis treatment due to medical history
11. Start of or planned start of an analgesic treatment or non-drug therapy, that significantly modulates pain perception, during trial participation
12. Planned surgery or other invasive procedure that requires analgetic treatment or might cause pain that could interfere with the low back pain intensity assessment
13. Patients with history of cancer in the last 5 years prior Visit 1. Except for cutaneous basal cell or squamous cell cancer resolved by excision without recurrence and cervical cancer in situ resolved by excision with negative pap test
14. Painful comorbidities which could interfere with the low back pain intensity assessment during the trial
15. Known history of human immunodeficiency virus (HIV) infection
16. Severe forms of the following diseases: anaemia, haematological/autoimmune/ endocrine/renal/hepatic/respiratory/cardiovascular/neurological/gastrointestinal/ symptomatic peripheral vascular diseases
17. Cardiovascular event in the last 3 months prior Visit 1
18. Poorly managed high blood pressure and/or untreated hypothyroidism
19. Patients with bilirubin metabolic disorder (e.g., Crigler-Najjar syndrome, Rotor syndrome)
20. Known history of major trauma or back surgery in the last 6 months prior Visit 1)
21. Known history of previous or current severe psychiatric illness Examples (not fully exhaustive) for severe psychiatric illness are: Bipolar (I or II) disorder, schizophrenia, manic episode, hypomanic episode, post-traumatic stress disorder, panic disorder, any psychotic disorder
22. Known history of previous or current severe depression (not due to chronic low back pain) and/or suicidal ideation at Visit 1
23. Known history of previous or current epilepsy or seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy based on pain reduction | End of the Treatment Phase (Week 7) compared to Baseline (Week -1)
  Change in mean pain intensity measured on an 11-point numerical rating scale (NRS)

SECONDARY OUTCOMES:
Pain responders | End of the Treatment Phase (Week 7) compared to Baseline (Week -1)
  Number and percentage of 30% and 50% pain responders
PGIC | At the end of the Treatment Phase (Week 7)
  Percentage of patients by answer category ('Improved', 'Not improved') of the global assessment of symptoms (PGIC, 7-point Likert scale where 0=very much better to 6=very much worse)
Safety: TEAEs and TESAEs | Week 1 up to Week 13
  Occurrence of treatment-emergent adverse events (TEAEs)/treatment-emergent serious adverse events (TESAEs)
Satisfaction with tolerability | At the end of the Treatment Phase (Week 7)
  Percentage of patients by answer category ("satisfied", "unsatisfied") based on the satisfaction of the patient with tolerability (5-point Likert scale, where 0=very satisfied to 4=very unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Johnson, Dr., Principal Investigator — St Pancras Clinical Research
Locations (1):
- St Pancras Clinical Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No